CLINICAL TRIAL: NCT04839042
Title: A Phase 1, First-In-Human, Open-label, Single Ascending Dose and Multidose Study to Assess the Safety, Reactogenicity, and Immunogenicity of the Adenovirus Vector SARS-CoV-2 Investigational Product SC-Ad6-1 Given Via Intramuscular, Intranasal or Inhaled Administration in Healthy Volunteers
Brief Title: A Phase 1, First-In-Human Study of the Investigational COVID-19 Vaccine SC-Ad6-1 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Moat Biotechnology Corporation (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: SC-Ad6-1-002
Record Dates: First submitted 2021-04-07; First posted 2021-04-09 (Actual); Last update posted 2025-08-21 (Actual); Status verified 2025-08

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (18):
- SC-Ad6-1 Low Dose Intramuscular (Experimental): Low Dose SC-Ad6-1, I.M., single-dose (Day 1)
  Interventions: Biological: SC-Ad6-1
- SC-Ad6-1 Medium Dose Intramuscular (Experimental): Medium Dose SC-Ad6-1, I.M., single-dose (Day 1)
  Interventions: Biological: SC-Ad6-1
- SC-Ad6-1 High Dose #1 Intramuscular (Experimental): High Dose #1 SC-Ad6-1, I.M., single-dose (Day 1)
  Interventions: Biological: SC-Ad6-1
- SC-Ad6-1 High Dose #2 Intramuscular (Experimental): High Dose #2 SC-Ad6-1, I.M., single-dose (Day 1)
  Interventions: Biological: SC-Ad6-1
- SC-Ad6-1 Multiple Dose Intramuscular (Experimental): Multiple Dose SC-Ad6-1, I.M., multiple-dose (Day 1 and Day 22)
  Interventions: Biological: SC-Ad6-1
- SC-Ad6-1 High Dose #3 Intramuscular Booster (Experimental): High Dose #3 SC-Ad6-1, I.M., single-dose booster (Day 1)
  Interventions: Biological: SC-Ad6-1
- SC-Ad6-1 Low Dose Intranasal (Experimental): Low Dose SC-Ad6-1, I.N., single-dose (Day 1)
  Interventions: Biological: SC-Ad6-1
- SC-Ad6-1 Medium Dose Intranasal (Experimental): Medium Dose SC-Ad6-1, I.N., single-dose (Day 1)
  Interventions: Biological: SC-Ad6-1
- SC-Ad6-1 High Dose #1 Intranasal (Experimental): High Dose #1 SC-Ad6-1, I.N., single-dose (Day 1)
  Interventions: Biological: SC-Ad6-1
- SC-Ad6-1 High Dose #2 Intranasal (Experimental): High Dose #2 SC-Ad6-1, I.N., single-dose (Day 1)
  Interventions: Biological: SC-Ad6-1
- SC-Ad6-1 Multiple Dose Intranasal (Experimental): Multiple Dose SC-Ad6-1, I.N., multiple-dose (Day 1 and Day 22)
  Interventions: Biological: SC-Ad6-1
- SC-Ad6-1 High Dose #3 Intranasal Booster (Experimental): High Dose #3 SC-Ad6-1, I.N., single-dose booster (Day 1)
  Interventions: Biological: SC-Ad6-1
- SC-Ad6-1 High Dose #4 Intranasal Booster (Experimental): High Dose #4 SC-Ad6-1, I.N., single-dose booster (Day 1)
  Interventions: Biological: SC-Ad6-1
- SC-Ad6-1 Low Dose Inhaled (Experimental): Low Dose SC-Ad6-1, I.H., single-dose booster (Day 1)
  Interventions: Biological: SC-Ad6-1
- SC-Ad6-1 Medium Dose Inhaled (Experimental): Medium Dose SC-Ad6-1, I.H., single-dose booster (Day 1)
  Interventions: Biological: SC-Ad6-1
- SC-Ad6-1 Multiple High Dose Intranasal (Experimental): Multiple High Dose SC-Ad6-1, I.N., multiple-dose (Day 1 and Day 29)
  Interventions: Biological: SC-Ad6-1
- SC-Ad6-1 Multiple High Dose Inhaled (Experimental): Multiple High Dose SC-Ad6-1, I.H., multiple-dose (Day 1 and Day 29)
  Interventions: Biological: SC-Ad6-1
- SC-Ad6-1 Multiple High Dose #2 Intranasal or Inhaled (Experimental): Multiple High Dose #2 SC-Ad6-1, I.N. or I.H., multiple-dose (Day 1 and Day 29)
  Interventions: Biological: SC-Ad6-1

INTERVENTIONS:
Biological: SC-Ad6-1 — SC-Ad6-1, I.M., single or multiple-dose
  Arms: SC-Ad6-1 High Dose #1 Intramuscular; SC-Ad6-1 High Dose #2 Intramuscular; SC-Ad6-1 High Dose #3 Intramuscular Booster; SC-Ad6-1 Low Dose Intramuscular; SC-Ad6-1 Medium Dose Intramuscular; SC-Ad6-1 Multiple Dose Intramuscular
Biological: SC-Ad6-1 — SC-Ad6-1, I.N., single or multiple-dose
  Arms: SC-Ad6-1 High Dose #1 Intranasal; SC-Ad6-1 High Dose #2 Intranasal; SC-Ad6-1 High Dose #3 Intranasal Booster; SC-Ad6-1 High Dose #4 Intranasal Booster; SC-Ad6-1 Low Dose Intranasal; SC-Ad6-1 Medium Dose Intranasal; SC-Ad6-1 Multiple Dose Intranasal; SC-Ad6-1 Multiple High Dose #2 Intranasal or Inhaled; SC-Ad6-1 Multiple High Dose Intranasal
Biological: SC-Ad6-1 — SC-Ad6-1, I.H., single or multiple-dose
  Arms: SC-Ad6-1 Low Dose Inhaled; SC-Ad6-1 Medium Dose Inhaled; SC-Ad6-1 Multiple High Dose #2 Intranasal or Inhaled; SC-Ad6-1 Multiple High Dose Inhaled

SUMMARY:
This is a single-centre, open-label, first-in-human, single ascending dose and multiple dose study to assess the safety, reactogenicity, and immunogenicity of the SC-Ad6-1 investigational product when administered via the intramuscular (IM), intranasal (IN) or inhaled (IH) route in healthy volunteers.

ELIGIBILITY:
Key Inclusion Criteria:

* Adult males and females, 18 to 60 years of age (inclusive)
* Body mass index ≥ 18.0 and ≤ 32.0 kg/m2, with a body weight ≥ 50 kg at screening
* Must have been fully vaccinated against COVID-19 and received last dose not less than 3 months prior to Day 1 (High Dose #3 I.M. and I.N. booster arms only), not less than 5 months prior to Day 1 (High Dose #4 I.N. booster arm only) and not less than 12 months prior to Day 1 (I.H. booster arms and I.N or I.H. multiple dose booster arms only)

Key Exclusion Criteria:

* History or presence of significant cardiovascular, pulmonary, hepatic, renal, haematological, gastrointestinal, endocrine, immunologic, dermatologic or neurological disease
* History of chronic respiratory disorders including asthma, emphysema, interstitial lung disease, pulmonary hypertension, recurrent pneumonia, or recent (≤14 days prior to Screening) or ongoing respiratory tract infection
* History of thrombosis (e.g., deep vein thrombosis, pulmonary embolism, etc.), any coagulation dysregulation disorder, or a history of thrombosis noted in immediate family members
* History of any neurological disorders or seizures including Guillain-Barre syndrome, with the exception of febrile seizures during childhood
* Known previous infection with SARS-CoV-2 or presence of antibodies against SARS-CoV-2 or a positive SARS-CoV-2 PCR test (non-booster arms only)
* Any history of malignant disease ≤5 years prior to registration
* History of clinically relevant immunosuppression from, but not limited to, immunodeficiency conditions such as common variable hypogammaglobulinemia

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 196 (Actual)
Dates: Start 2021-06-28 (Actual); Primary Completion 2025-03-04 (Actual); Study Completion 2025-03-04 (Actual)

PRIMARY OUTCOMES:
Number of participants with solicited local and systemic adverse events for 7 days Following Each Dose | 7 days following each dose
  Solicited local adverse events are defined as pain, redness and swelling at the site of dose administration for the intramuscular arms, are defined as stuffy nose, runny nose, nasal discomfort, loss of smell, sore or scratchy throat for the intranasal arms and are defined as stuffy nose, runny nose, dry mouth, mouth sores, sore or scratchy throat and cough for the inhalation arms. Solicited systemic adverse events for all routes of administration are defined as fever, headache, muscle pain, joint pain, fatigue, nausea or vomiting, and chills.
Incidence and severity of adverse events (AEs), including withdrawals due to safety or tolerability reasons | Up to 106 days following first dose
Humoral response to SARS-CoV-2 as measured by neutralizing antibodies using wild-type virus assay | Up to 106 days following first dose

SECONDARY OUTCOMES:
Humoral response to SARS-CoV-2 as measured by serum IgG and IgA antibodies to the SARS-CoV-2 spike protein (ELISA) | Up to 106 days following first dose
Humoral response to SARS-CoV-2 as measured by mucosal IgA antibodies to the SARS-CoV-2 spike protein (ELISA) and total mucosal IgA | Up to 106 days following first dose
Measurement of cytokine-producing T cells specific for the SARS-CoV-2 spike protein (ELISpot) | Up to 106 days following first dose
Measurement of adenovirus 6 (Ad6) neutralizing antibodies (anti-drug antibodies (ADA)) | Up to 106 days following first dose

CONTACTS AND LOCATIONS:
Overall Officials: Russell Rother, Ph.D., Study Director — Moat Biotechnology Corporation
Locations (1):
- Tetherex Study Site, Brisbane, Queensland, Australia

IPD SHARING:
Plan to Share IPD: No